CLINICAL TRIAL: NCT02732678
Title: Dose-Finding of Propranolol in Combination With Metronomic Fixed Oral Cyclophosphamide Based on Bivariate Efficacy-tolerability Outcome in Patients With Locally Advanced or Metastatic Angiosarcoma: A Collaborative and Innovative Phase I-II Sequential Trial by the French Sarcoma Group (GSF/GETO)
Acronym: PROPAN
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2015-005177-21; 2015-29 (Other: AP-HM)
Record Dates: First submitted 2016-03-29; First posted 2016-04-11 (Estimated); Last update posted 2016-04-11 (Estimated); Status verified 2016-04

CONDITIONS: Angiosarcoma
MeSH Terms: conditions — Hemangiosarcoma | interventions — Propranolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort of a dose of Propranolol 80 mg/day (Experimental)
  Interventions: Drug: PROPRANOLOL
- Cohort of a dose of Propranolol 120 mg/day (Experimental)
  Interventions: Drug: PROPRANOLOL
- Cohort of a dose of Propranolol 160 mg/day (Experimental)
  Interventions: Drug: PROPRANOLOL

INTERVENTIONS:
Drug: PROPRANOLOL

SUMMARY:
Adrenergic processes stimulated by epinephrine and norepinephrine drive to the development of tumor growth and metastasis. Beta-adrenergic receptor (BAR) antagonists have shown efficacy against melanoma, breast cancer and prostate cancer. The non-specific BAR inhibitor propranolol has been used as the gold standard treatment in pediatric patients with benign infantile hemangioma which express high levels of beta adrenergic receptors potentially explaining their sensitively to propranolol. BAR have been shown to be expressed across a diverse panel of vascular tumors, with the highest expression in malignant vascular tumors including angiosarcoma. Several reports indicate positive results from beta-blockade in patients with moderately threatening vascular tumors. It remains to be determined if more malignant vascular tumor such as the angiosarcomas are susceptible to propranolol. Besides, due to the lack of adequate therapies for angiosarcoma (doxorubicin or paclitaxel and finally cyclophosphamide in third line) and to the poor prognosis of this rare and aggressive tumor, there is a strong need for the development of treatments against this tumor type. Recently using a panel of angiosarcoma cell lines. demonstrate that beta-adrenergic inhibition blocks cell proliferation and induces apoptosis in a dose dependent manner. Moreover, using in vivo tumor models they demonstrate that propanolol shows remarkable efficacy in reducing the growth of angiosarcoma tumors. Based on these proofs of mechanisms in vitro and in vivo and due to the well established safety propranolol in humans, investigators propose to determine among a wide range of propranolol dose (80 mg/d ; 120 mg/d and 160 mg/d) the optimal one based on bivariate efficacy-toxicity outcome in patients with angiosarcoma treated by cyclophosphamide. Because these two drugs have different pharmacological mechanisms, the aim is to determine the optimal dose of propranolol having the best systemic cardiovascular tolerability and the best potential antiangiogenic effect in addition with cyclophosphamide.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent > 15 years with a body surface >1,6 m2
* Histologically proven angiosarcoma, reviewed by an independent pathologist, with metastasis or locally advanced stage not amenable to radiotherapy or curative-intent surgery after multidisciplinary decision ;
* Prior systemic treatment with paclitaxel or doxorubicin
* At least one lesion measurable according to the RECIST, version 1.1;
* No brain or meningeal metastasis;
* No more than two prior lines of chemotherapy (whatever the indication);
* A World Health Organization performance status score ≤2;
* Neutrophils count > 1000 /mm3, platelets count ≥100,000/mm3, hemoglobin level ≥ 8 g/Dl, liver transaminases ≤1.5 XULN, total bilirubin ≤1.5X ULN, serum creatinine≤1.5XULN, and amylase and lipase≤1.5XULN

Exclusion Criteria:

* Pregnant or breast-feeding women.
* Subject with a contraindication to propranolol (ie cardiogenic shock; sinus bradycardia and greater than first-degree block; Chronic Obstructive Pulmonary Disease and bronchial asthma; patients with known hypersensitivity to Propranolol; assessed by cardiovascular and pulmonary history and examinations including blood pressure, ECG; untreated Pheochromocytoma, Congestive heart failure not controlled by treatment, Prinzmetal's angina)
* Subject with Severe Raynaud Phenomena or Raynaud Disease
* Subject with Prior systemic treatment with Cyclophosphamide as 1st or 2nd line

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2016-05; Primary Completion 2018-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
toxicity of each tested propranolol dose level in association to cyclophosphamide assessed according to NCI-CTC AE Version 4.0 | 1 month
  The toxicity of propranolol is well described on humans as well as its pharmacokinetic (Peak plasma concentrations occur about 1 to 4 hours) after oral dose and pharmacodynamics characteristics with the main target on beta-adrenergic receptor (blocking agent possessing no other autonomic nervous system activity). In this study the toxicity of each tested propranolol dose level in association to cyclophosphamide will be assessed according to NCI-CTC AE Version 4.0 at 1 month (Recording AE, Blood pressure, and electrocardiography). A dose-limiting toxicity (DLT) will be considered as any grade 3 or higher specially cardiac and hematologic but also non-hematologic toxicity that is probably or definitely related to treatment.
Non-progression rate | 3 month
  The efficacy criterion is defined as the non-progression rate at 3 months according to RECIST 1.1 guidelines and with central radiological review.

CONTACTS AND LOCATIONS:
Overall Officials: Urielle Desalbres, Study Director — Assistance Publique Hôpitaux de Marseille; Sébatien SALAS, MD PhD, Principal Investigator — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseill, France

IPD SHARING:
Plan to Share IPD: No